CLINICAL TRIAL: NCT00859287
Title: Omepral® Tablets Mega-study to Investigate the Efficacy on Various Type of Acid Reflux Related Symptoms and QOL, and Epidemiology in Patients With Erosive Esophagitis in Daily Medical Practice
Brief Title: Omepral® Tablets Special Clinical Experience Investigation in Patients With Erosive Esophagitis
Acronym: OMAREE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Huvenne, Alain / Senior Medical Marketing Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-GJP-DUM-2007/1
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Reflux Esophagitis
Keywords: Reflux esophagitis; Omepral®; QOLRAD
MeSH Terms: conditions — Esophagitis, Peptic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This open label, non-interventional study is to compare the efficacy of Omepral® tablet and any other treatments excepting proton pump inhibitors (PPIs) for the treatment of various type of acid reflux related symptoms in patients with reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed as erosive esophagitis or history of erosive esophagitis confirmed by endoscopy.
* Patients who answered questionnaires of quality of life (QOLRAD-J), symptom severity and frequency and treatment satisfaction.
* During the past 1 week , patients who have either two days or more with heartburn or acid taste in the mouth of any severity

Exclusion Criteria:

* Patients receiving treatment with proton pump inhibitors, which make stomach acid decreased during the last 4 weeks prior to enrolment.
* Patients who cannot answer questionnaires of quality of life (QOLRAD-J), symptom severity and frequency and treatment satisfaction.
* Patients included previously in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients endoscopically diagnosed as erosive esophagitis accompanied with either two days or more heartburn or acid taste in the mouth of any severity
Sampling Method: Non-Probability Sample
Enrollment: 10703 (Actual)
Dates: Start 2007-06; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Patients symptom evaluated by investigator | at entry, 4 weeks and 8 weeks
Patients reported symptom | at entry, 4 weeks and 8 weeks

SECONDARY OUTCOMES:
Patients reported outcome score | at entry, 4 weeks and 8 weeks
Adverse event | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Japan Medical Director MD, Study Director — AstraZeneca

REFERENCES:
- [Derived] Yoshida S, Nii M, Date M. Effects of omeprazole on symptoms and quality of life in Japanese patients with reflux esophagitis: final results of OMAREE, a large-scale clinical experience investigation. BMC Gastroenterol. 2011 Feb 28;11:15. doi: 10.1186/1471-230X-11-15. PMID 21356058